CLINICAL TRIAL: NCT02195986
Title: Clinical Endpoint Therapeutic Equivalence Multi-Site Study Comparing Estradiol Vaginal Cream (0.01%; Mylan) to Estrace® Cream (0.01%; Warner Chilcott) in Postmenopausal Females With Atrophic Vaginitis
Brief Title: A Comparison of Estradiol Vaginal Cream to Estrace® Cream in 350 Postmenopausal Females With Atrophic Vaginitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVCR-11196
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Results first posted 2017-09-06 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Atrophic Vaginitis
Keywords: vaginal dryness; vaginal and/or vulvar irritation/itching; dysuria; vaginal pain and bleeding associated with sexual activity; vaginal atrophy
MeSH Terms: conditions — Atrophic Vaginitis; Pruritus; Dysuria | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estradiol Vaginal Cream (Experimental): Estradiol Vaginal Cream, 0.01%, administered once daily for 7 days.
  Interventions: Drug: Estradiol Vaginal Cream, 0.01%
- Estrace® 0.01% cream (Active Comparator): Estrace® 0.01% vaginal cream, administered once daily for 7 days.
  Interventions: Drug: Estrace® 0.01% cream
- Placebo Vaginal Cream (Placebo Comparator): Placebo Vaginal Cream, administered once daily for 7 days.
  Interventions: Drug: Placebo Vaginal Cream

INTERVENTIONS:
Drug: Estradiol Vaginal Cream, 0.01% — Estradiol Vaginal Cream, 0.01% (1 x 2g for 7 days)
  Arms: Estradiol Vaginal Cream
Drug: Estrace® 0.01% cream — Estrace® 0.01% vaginal cream ( 1 x 2g for 7 days)
  Arms: Estrace® 0.01% cream
Drug: Placebo Vaginal Cream — Placebo Vaginal Cream ( 1 x 2 g for 7 days)
  Arms: Placebo Vaginal Cream

SUMMARY:
The purpose of this study is to determine the therapeutic equivalence of Mylan's estradiol vaginal cream to Estrace® cream and superiority of both products to placebo. The protocol describes a randomized, double-blind, multi-dose, placebo-controlled, parallel study of a 7 day treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of providing informed consent.
2. Age: 40-70 years old.
3. Sex: Female
4. Postmenopausal defined as at least 12 months of spontaneous amenorrhea or at least 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/ml or at least 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
5. Weight: At least 48 kg with all subjects having a Body Mass Index less than or equal to 38 kg/m2 but greater than or equal to 19 kg/m2.
6. Baseline evaluation requirements:

   * ≤5% superficial cells on vaginal smear cytology
   * Vaginal pH > 5.0
   * At least one patient self-assessed moderate to severe symptom of vulvar and/or vaginal atrophy (VVA) from the following list that is identified by the subject:
   * Vaginal dryness
   * Vaginal and/or vulvar irritation/itching
   * Dysuria
   * Vaginal pain associated with sexual activity
   * Vaginal bleeding associated with sexual activity (absence vs. presence)
7. All subjects should be judged to be eligible for participation in this study by the principal or sub-investigator physician during a pre-study medical evaluation performed within 28 days of the initial dose of study medication which will include:

   1. a normal or non-clinically significant physical examination, including vital signs
   2. a normal or non-clinically significant pelvic examination that was consistent with hypoestrogenemia
   3. a normal or non-clinically significant breast exam and mammogram
   4. a normal or non-clinically significant ASCUS Papanicolaou ("Pap") smear that is negative for HPV for subjects with an intact uterus and cervix
   5. within normal limits or non-clinically significant laboratory evaluation results (unless otherwise noted in the exclusion criteria) for the following tests:

      * Serum Chemistry
      * Hematology
      * Coagulogram
      * Urinalysis
   6. normal or non-clinically significant 12- Lead ECG.
   7. negative urine drug screen including amphetamine, barbiturates, benzodiazepines, cannabinoid, cocaine, opiates, methadone and phencyclidine with the following exceptions: positive tests for amphetamines, barbiturates, benzodiazepines, or opiates may be allowed provided the subject has a valid prescription and is on a stable regimen that complies with Exclusion Criteria, Section 6.3.2.
   8. negative urine cotinine test.
8. For women with an intact uterus, an endometrial thickness < 5 mm as determined by vaginal ultrasonography.
9. If warranted, other tests or examinations may be performed at the discretion of the Principal Investigator or responsible physician.
10. Ability to use applicator properly.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Any contraindication to estrogen therapy.
3. Social Habits:

   1. Use of any tobacco-containing products within 1 year of the start of the study.
   2. Regular intake of more than 7 units of alcohol per week.
   3. Beginning any new regimens of vitamins or herbal products within 7 days prior to the initial dose of the study medication.
   4. Any recent, significant change in dietary or exercise habits.
   5. History of drug and/or alcohol abuse within one year of start of study.
4. Medications:

   1. Use of any new prescription or over-the-counter (OTC) medication regimens within fourteen (14) days prior to the initial dose of study medication (any necessary medication, unless otherwise noted in the exclusion criteria, for which dosing has been stabilized for a period of at least 14 days prior to initial dosing of study drug and is expected to remain stable for the entire study period is allowed, with the exception of acetaminophen, which may be administered as needed to treat minor adverse events).
   2. Use of hormonal replacement therapies for the following time periods:

      * within 2 weeks of baseline assessment for vaginal therapy (rings, creams, gels)
      * within 4 weeks of baseline assessment for transdermal estrogen alone or estrogen/progestin therapy
      * within 8 weeks of baseline assessment for oral estrogen and/or progestin therapy or intrauterine progestin therapy
      * within 3 months of baseline assessments for progestin implants or estrogen alone injectable therapy
      * within 6 months of baseline assessments for estrogen pellet or progestin injectable therapy
   3. A depot injection or implant of any drug within 3 months prior to administration of study medication.
   4. Currently taking medication indicated for anticoagulation as a result of an excluded condition listed in #5 below. This includes but is not limited to warfarin, heparin, NSAIDs, clopidogrel, dabigatran, etc.
5. Diseases:

   1. History of any significant cardiovascular, hepatic, renal, pulmonary, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, psychological, urinary, musculoskeletal disease or malignancies unless under medical control and/or deemed not clinically significant by the Principal Investigator or Medical Sub-investigator.
   2. Manifestation or treatment for significant cardiovascular disease (congestive heart failure, stroke or ischemic attack, myocardial infarction, coronary artery bypass, percutaneous angioplasty or > 50% angiographic narrowing of coronary artery, thrombosis of deep veins and arteries, thromboembolic disorders, pulmonary embolism) or history of these conditions.
   3. Coronary artery or cerebrovascular disease.
   4. Current clinically significant liver or kidney dysfunction/disorders.
   5. Current clinically significant gallbladder dysfunction/disorders.
   6. Abnormal or clinically significant breast examination. Acceptable breast examination is defined as no masses or other findings identified that are suspicious of malignancy.
   7. First degree family history of breast cancer.
   8. Current non diet controlled diabetes mellitus or other clinically significant endocrinological disease.
   9. Estrogen-dependent neoplasia
   10. Postmenopausal uterine bleeding
   11. Endometrial hyperplasia
   12. Uncontrolled hypothyroidism
   13. Urinalysis showing an ongoing clinically significant urinary tract infection that requires treatment.
   14. Current clinically significant vaginal infection that requires treatment.
   15. Known chronic lichen sclerosis
   16. Acute illness at the time of either the pre-study medical evaluation or dosing.
   17. History of allergy or hypersensitivity to estradiol, other related products, or any inactive ingredients.
   18. Undiagnosed vaginal bleeding or history of significant risk factors for endometrial cancer.
   19. Increased frequency or severity of headaches while on previous hormone or estrogen therapy.
   20. History of psychiatric disorders occurring within the last 6 months that require hospitalization or medication.
   21. Current hypercalcemia, hypocalcemia, and/or hypertriglyceridemia.
   22. Clinically significant eye/visual abnormalities such as retinal vascular thrombosis, partial or complete loss of vision, proptosis, diplopia, papilledema, retinal vascular lesions.
6. Any reason which, in the opinion of the Principal Investigator or Medical Sub-Investigator, would prevent the subject from safely participating in the study.
7. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.
8. Sitting blood pressure higher than 150/90 mmHg at screening.
9. Baseline serum estradiol levels >30 pg/mL at screening.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Hummel, Ph.D., Study Chair — Mylan Pharmaceuticals Inc; Ronald Ackerman, M.D., Principal Investigator — Comprehensive Clinical Trials, LLC; James Andersen, M.D., Principal Investigator — Meridien Research; Keith Aqua, M.D., Principal Investigator — Visions Clinical Research; Theodore Cooper, M.D., Principal Investigator — Horizons Clinical Research Center, LLC; Scott Eder, M.D., Principal Investigator — Women's Health Research Center/The Center for Women's Health & Wellness, LLC; William Koltun, M.D., Principal Investigator — Medical Center for Clinical Research; Gigi Lefebvre, M.D., Principal Investigator — Meridien Research; Leonard Ranasinghe, M.D., Principal Investigator — Northern CA Research; Rovena Reagan, M.D., Principal Investigator — Women's Health Care Research Corp.; Ronald Surowitz, D.O., Principal Investigator — Health Awareness, Inc.; Steven Sussman, M.D., Principal Investigator — Lawrence OB/GYN Clinical Research, LLC; G. Michael Swor, M.D., Principal Investigator — Physician Care Clinical Research LLC; Olga Tudela, M.D., Principal Investigator — Veritas Research., Corp.; Arthur Waldbaum, M.D., Principal Investigator — Downtown Women's Health Care; Maria C Fernandez, M.D., Principal Investigator — South Coast Research Center, Inc.; Gary Carson, M.D, Principal Investigator — Northern CA Research; Lydie Hazan, M.D., Principal Investigator — Axis Clinical Trials; Alfred Moffett, M.D., Principal Investigator — OB-GYN Associates of Mid Florida; Tracey Lemon, M.D., Principal Investigator — Georgia Center for Women; Steven Foley, M.D., Principal Investigator — MCB Clinical Research Centers, LLC; Jason Haffizulla, M.D., Principal Investigator — Sunrise Medical Research, Inc.; Robert Hunter, M.D., Principal Investigator — ARA-Arizona Research Associates
Locations (21):
- United States (21):
  - ARA-Arizona Research Associates, Tucson, Arizona
  - Axis Clinical Trials, Los Angeles, California
  - Northern CA Research, Sacramento, California
  - MCCR, San Diego, California
  - Women's Health Care Research Corp., San Diego, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Downtown Women's Health Care, Denver, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Sunrise Medical Research, Coral Springs, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Meridien Research, Lakeland, Florida
  - OB-GYN Associates of Mid Florida, Leesburg, Florida
  - SouthCoast Research Center, Miami, Florida
  - Veritas Research, Corp., Miami Lakes, Florida
  - Physician Care Clinical Research LLC, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Sunrise Medical Research, Tamarac, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Georgia Center for Women, Atlanta, Georgia
  - Lawrence OB/GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Women's Health Research Center/The Center for Women's Health & Wellness, LLC, Plainsboro, New Jersey

IPD SHARING:
Plan to Share IPD: No
N/A - Phase I study

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol Vaginal Cream: Estradiol Vaginal Cream, 0.01%, administered once daily for 7 days.
  Estradiol Vaginal Cream, 0.01%: Estradiol Vaginal Cream, 0.01% (1 x 2 g for 7 days)
- Estrace® 0.01% Cream: Estrace® 0.01% vaginal cream, administered once daily for 7 days.
  Estrace® 0.01% cream: Estrace® 0.01% vaginal cream (1 x 2 g for 7 days)
- Placebo Vaginal Cream: Placebo Vaginal Cream, administered once daily for 7 days.
  Placebo Vaginal Cream: Placebo Vaginal Cream (1 x 2 g for 7 days)
Period: Overall Study
Arm/Group | Estradiol Vaginal Cream | Estrace® 0.01% Cream | Placebo Vaginal Cream
Started | 146 | 147 | 73
Completed | 143 | 142 | 71
Not Completed | 3 | 5 | 2
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Family Emergency | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Non-compliance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes all randomized subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Estradiol Vaginal Cream | Estrace® 0.01% Cream | Placebo Vaginal Cream | Total
Number analyzed (Participants) | 146 | 147 | 73 | 366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 128 | 124 | 61 | 313
  >=65 years | 18 | 23 | 12 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (5.25) | 59.6 (5.88) | 59.4 (5.82) | 59.4 (5.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 147 | 73 | 366
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 23 | 13 | 66
  Not Hispanic or Latino | 116 | 124 | 60 | 300
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 18 | 11 | 44
  White | 130 | 125 | 61 | 316
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 146 | 147 | 73 | 366
Height [Mean (Standard Deviation); unit: cm] | 162.1 (6.43) | 161.5 (6.18) | 162.6 (6.55) | 161.9 (6.35)
Weight [Mean (Standard Deviation); unit: kg] | 69.77 (12.74) | 69.39 (12.67) | 67.61 (11.37) | 69.19 (12.44)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (4.41) | 26.6 (4.56) | 25.6 (4.11) | 26.4 (4.42)

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint (Vaginal Cytology + Vaginal pH) Equivalence
Description: Treatment comparison of the proportion of patients in the Per Protocol (PP) population who received either Estradiol Vaginal Cream or Estrace® that were identified as responders at the end of the treatment period on Study Day 8.
  A responder was defined as a patient with at least a 25% reduction from baseline in the sum of % basal/parabasal + % intermediate cells on vaginal cytology AND vaginal pH ≤ 5.0 with a change from baseline vaginal pH of at least 0.5.
Time Frame: Study Day 8
Population: The Per Protocol population was used for the primary endpoint equivalence comparison which consisted of all randomized subjects that were dosed with 75%-125% of scheduled applications of Test or Reference and completed primary endpoint evaluation on Study Day 8 +/- 2 days with no protocol violations that would affect treatment evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol Vaginal Cream | Estrace® 0.01% Cream
Number analyzed (Participants) | 111 | 117
Participants | 42 | 45
Statistical Analysis 1: Comparison: Estradiol Vaginal Cream vs Estrace® 0.01% Cream; The compound hypothesis to test was: H0: PT -PR < -.20 or PT -PR > .20 versus HA : -.20 ≤ PT -PR ≤ .20 Where PT = cure rate of test treatment, and PR = cure rate of reference treatment; Test type: Equivalence — Bioequivalence was established for the primary endpoint if the 90% confidence interval for the difference of responder rates (test - reference) from baseline to Day 8 for the primary endpoint is contained within [-0.20, 0.20], using the per-protocol population; Difference = -0.0062, 90% CI 2-sided [-0.1209 to 0.1084]

2. Primary Outcome: Primary Endpoint (Vaginal Cytology + Vaginal pH) Comparison of Active Treatments to Placebo
Description: Treatment comparison of the proportion of patients in the Per Protocol (PP) population who received either Estradiol Vaginal Cream, Estrace®, or Placebo that were identified as responders at the end of the treatment period on Study Day 8.
  A responder was defined as a patient with at least a 25% reduction from baseline in the sum of % basal/parabasal + % intermediate cells on vaginal cytology AND vaginal pH ≤ 5.0 with a change from baseline vaginal pH of at least 0.5.
Time Frame: Study Day 8
Population: The Intent-to-treat (ITT) population was used for the comparison of active treatments versus placebo analysis which consisted of all randomized subjects that used at least one dose of Test, Reference or Placebo and returned for at least one post-baseline visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol Vaginal Cream | Estrace® 0.01% Cream | Placebo Vaginal Cream
Number analyzed (Participants) | 125 | 138 | 65
Participants | 49 | 51 | 1
Statistical Analysis 1: Comparison: Estradiol Vaginal Cream vs Placebo Vaginal Cream; Both the test and reference products should both be statistically superior to placebo (p<0.05, two-sided) using the Chi squared test with Yate's correction for the primary endpoint responder rate, using the ITT study population and last observation carried forward. The compound hypothesis to test was: H0: PT - PP ≤ 0 versus HA: PT - PP > 0; Where PT = cure rate of test treatment, and PP = cure rate of placebo; Test type: Superiority — Superiority test of test product vs placebo; p < 0.0001, Chi-squared; Difference = 0.3766, 95% CI 2-sided [0.2743 to 0.4790]
Statistical Analysis 2: Comparison: Estrace® 0.01% Cream vs Placebo Vaginal Cream; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Superiority test of reference product vs placebo; p < 0.0001, Chi-squared; Difference = 0.3542, 95% CI 2-sided [0.2570 to 0.4514]

3. Secondary Outcome: Comparison of the Number of Participants With Treatment Success for the Patient Self-assessment of the Symptoms of Vulvar and Vaginal Atrophy - Equivalence
Description: Evaluation and comparison between Estradiol Vaginal Cream and Estrace® treatment groups of the change from baseline in the most bothersome vulvar and/or vaginal atrophy symptom including vaginal dryness, vaginal and/or vulvar irritation/itching, dysuria, vaginal pain associated with sexual activity, or vaginal bleeding associated with sexual activity as identified by each subject. A score ≤ 1 on Study Day 8 for the most bothersome symptom as identified by the subject at baseline (Study Day -1) was considered a treatment success. A score ≥ 2 on Study Day 8 for the most bothersome symptom as identified by the subject at baseline (Study Day -1) was considered a treatment failure.
Time Frame: Day 8
Population: The Per Protocol population was used for the secondary endpoint equivalence comparison which consisted of all randomized subjects that were dosed with 75%-125% of scheduled applications of Test or Reference and completed secondary endpoint evaluation on Study Day 8 +/- 2 days with no protocol violations that would affect treatment evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol Vaginal Cream | Estrace® 0.01% Cream
Number analyzed (Participants) | 97 | 91
Participants | 72 | 63
Statistical Analysis 1: Comparison: Estradiol Vaginal Cream vs Estrace® 0.01% Cream; Test type: Equivalence — Bioequivalence was established for the secondary endpoint if the 90% confidence interval for the difference of responder rates (test - reference) from baseline to Day 8 for the secondary endpoint is contained within [-0.20, 0.20], using the per-protocol population; Difference = 0.0500, 90% CI 2-sided [-0.0687 to 0.1686]

4. Secondary Outcome: Comparison of the Number of Participants With Treatment Success for the Patient Self-assessment of the Symptoms of Vulvar and Vaginal Atrophy - Comparison to Placebo
Description: Evaluation and comparison between Estradiol Vaginal Cream, Estrace®, and Placebo treatment groups of the change from baseline in the most bothersome vulvar and/or vaginal atrophy symptom including vaginal dryness, vaginal and/or vulvar irritation/itching, dysuria, vaginal pain associated with sexual activity, or vaginal bleeding associated with sexual activity as identified by each subject. A score ≤ 1 on Study Day 8 for the most bothersome symptom as identified by the subject at baseline (Study Day -1) was considered a treatment success. A score ≥ 2 on Study Day 8 for the most bothersome symptom as identified by the subject at baseline (Study Day -1) was considered a treatment failure.
Time Frame: Day 8
Population: The Intent-to-treat (ITT) population was used for the Superiority Analysis which consisted of all randomized subjects that used at least one dose of Estradiol Vaginal Cream, Estrace®, or Placebo and returned for at least one post-baseline visit
Measure: Count of Participants; unit: Participants
Arm/Group | Estradiol Vaginal Cream | Estrace® 0.01% Cream | Placebo Vaginal Cream
Number analyzed (Participants) | 111 | 107 | 55
Participants | 82 | 77 | 33
Statistical Analysis 1: Comparison: Estradiol Vaginal Cream vs Placebo Vaginal Cream; Both the test and reference products should both be statistically superior to placebo (p<0.05, two-sided) using the Chi squared test with Yate's correction for the secondary endpoint responder rate, using the ITT study population and last observation carried forward. The compound hypothesis to test was: H0: PT - PP ≤ 0 versus HA: PT - PP > 0; Where PT = cure rate of test treatment, and PP = cure rate of placebo; Test type: Superiority — Superiority test of test product vs placebo; p = 0.1092, Chi-squared; Difference = 0.1387, 95% CI 2-sided [-0.0280 to 0.3054]
Statistical Analysis 2: Comparison: Estrace® 0.01% Cream vs Placebo Vaginal Cream; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — Superiority test of reference product vs placebo; p = 0.1805, Chi-squared; Difference = 0.1196, 95% CI 2-sided [-0.0491 to 0.2883]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from signing of the ICF until 30 days post study exit on Study Day 8.
Description: Adverse events were collected via subject self-reporting in a diary and queries at clinic visits. Only subjects that were confirmed to have received at least 1 dose of study medication were included in the Safety Population (i.e., At risk) for adverse event reporting. The Safety Population consisted of 146 subjects for the Estradiol Vaginal Cream arm, 144 subjects for the Estrace® arm, and 72 subjects for the Placebo arm.
Arm/Group | Estradiol Vaginal Cream | Estrace® 0.01% Cream | Placebo Vaginal Cream
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/144 | 0/72
Serious Adverse Events (participants affected / at risk) | 1/146 | 0/144 | 0/72
Other Adverse Events (participants affected / at risk) | 31/146 | 27/144 | 8/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Vaginal Cream (N=146) | Estrace® 0.01% Cream (N=144) | Placebo Vaginal Cream (N=72)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial Haemorrhage (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol Vaginal Cream (N=146) | Estrace® 0.01% Cream (N=144) | Placebo Vaginal Cream (N=72)
Abdominal Pain (Gastrointestinal disorders) | 12 (13) | 17 (22) | 0 (0)
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 9 (10) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 9 (11) | 4 (4) | 4 (4)
Breast Tenderness (Reproductive system and breast disorders) | 2 (2) | 8 (8) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes